CLINICAL TRIAL: NCT06578624
Title: A Phase 1/2a, Open-Label Study of Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SA53-OS, an MDM2 Inhibitor, in Patients With Locally Advanced or Metastatic p53 Wild-Type Solid Tumors
Brief Title: Safety and Preliminary Efficacy of SA53-OS in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lamassu Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB-SA53-101
Record Dates: First submitted 2024-08-15; First posted 2024-08-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
Keywords: p53 wild-type tumor; liposarcoma; MDM2 inhibitor; solid tumors; dedifferentiated liposarcoma (DD LPS); p53; Advanced or metastatic solid tumors
MeSH Terms: conditions — Liposarcoma | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Phase 1 of the study will start with dose escalation by 2-fold (i.e., 2x preceding dose level) in cohorts of a single participant until Grade 2 or greater toxicity is observed. When a single Grade 2 or higher toxicity is observed, 3+3 multi-participant cohorts will be treated at the dose in which the Grade 2 or higher toxicity was observed by enrolling another 2 participants at this dose. The 3+3 multi-participant cohorts will follow the standard 3+3 paradigm based on occurrence of any DLT with 50% dose escalation until the MTD is identified. In phase 2 of the study, the MTD will be administered to 2 cohorts of 20 participants each: Cohort A) with known MDM2 amplified DD LPS; Cohort B) p53 wild-type solid tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Dose escalation phase
  Interventions: Drug: SA53-OS (phase 1)
- Phase 2 (Experimental): Cohort A: DDLPS (MDM2 amplified and p53 wild-type) Cohort B: other p53 wild-type solid tumors
  Interventions: Drug: SA53-OS (phase 2)

INTERVENTIONS:
Drug: SA53-OS (phase 1) — Dose escalation phase in which participants receive SA53-OS on 3 consecutive days every 3 weeks for a maximum of 2 years. Single participant cohorts will be enrolled until a Grade 2 or greater toxicity is observed and then 3+3 multi-participant cohorts will be enrolled until the MTD is identified.
  Arms: Phase 1
Drug: SA53-OS (phase 2) — Dose expansion phase in which participants receive SA53-OS on 3 consecutive days every 3 weeks for a maximum of 2 years at the MTD identified in phase 1.
  Arms: Phase 2

SUMMARY:
The objective of this study is to assess the safety, efficacy, and pharmacokinetics of SA53-OS in adult participants with refractory solid tumors.

The study is comprised of 2 parts: Part 1 called dose escalation, and Part 2a called dose expansion. This study starts with Part 1 where participants who are diagnosed with advanced or metastatic solid tumor cancers receive different doses of SA53-OS (starting with the lowest dose) to find the maximum tolerated dose (MTD) of SA53-OS. Once the MTD of SA53-OS is known, the study continues to Part 2a where participants who are diagnosed with dedifferentiated liposarcoma (DD LPS) or other solid tumor cancers will receive SA53-OS at the MTD.

The study drug, SA53-OS, will be administered for 3 consecutive days every 3 weeks as an oral solution for up to 2 years.

DETAILED DESCRIPTION:
This is a phase 1/2a, open-label, dose escalation study conducted in adult participants with p53 wild-type refractory solid tumors. The study will assess the safety, efficacy, and pharmacokinetics of SA53-OS a novel MDM2 inhibitor capable of selective activation of p53. This enables the p53 tumor suppressor protein to selectively facilitate tumor cell death and growth inhibition.

The study drug, SA53-OS, will be administered for 3 consecutive days every 3 weeks as an oral solution. Phase 1 will consist of a dose escalation study to establish a candidate recommended phase 2 dose (RP2D). Phase 2a will enroll 2 expansion cohorts to establish any preliminary efficacy of SA53-OS in participants with dedifferentiated liposarcoma (DD LPS) with MDM2 amplifications and other p53 wild-type solid tumors as a single agent.

Phase 1 dose escalation:

Escalating doses of SA53-OS will be provided to participants with p53 wild-type refractory solid tumors to determine the RP2D. The MTD is the highest dose of a drug or treatment that does not cause unacceptable side effects in the first cycle. The RP2D considers all available safety, pharmacokinetics, and efficacy data including, the frequency, severity, and manageability of toxicities occurring after Cycle 1.

Phase 1 of the study will start with dose escalation by 2-fold (i.e., 2x preceding dose level) in cohorts of a single participant until Grade 2 or greater toxicity is observed.

When a single Grade 2 or higher toxicity is observed, 3+3 multi-participant cohorts will be treated at the dose in which the Grade 2 or higher toxicity was observed by enrolling another 2 participants at this dose. The 3+3 multi-participant cohorts will follow the standard 3+3 paradigm based on occurrence of any DLT with 50% dose escalation until the MTD is identified.

Phase 2a dose expansion:

The purpose of Phase 2a of the study is to describe any preliminary evidence of efficacy from SA53-OS monotherapy in participants with DD LPS or other p53 wild-type or MDM2 amplified solid tumors. Phase 2a will also be used to confirm the safety and tolerability of the candidate RP2D of SA53-OS determined in Phase 1 of the study, to further describe the toxicity and pharmacokinetics profiles of SA53-OS, and to assess potential biomarkers of sensitivity resistance, and toxicity.

Participants will continue to receive study treatment until either: 1) disease progression; 2) occurrence of unacceptable treatment-related toxicity as per participant or Investigator discretion; 3) the maximum of 2 years of treatment has been reached; or 4) other reason(s) for study treatment discontinuation. In the case of complete response, treatment should be continued for at least 6 months if no other stopping criteria are met, and further treatment can be recommended at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Tumor characteristics of participants in Phase 1

  1. Histologically and/or cytologically confirmed diagnosis of advanced or metastatic solid tumor and/or non-Hodgkin lymphoma excluding primary central nervous system malignancy for which no standard effective treatment exists or where that treatment was declined. Participants with non-Hodgkin lymphoma should have failed ≥ 2 prior lines of systemic therapy prior enrollment.
  2. Tumor p53 wild-type.
* Tumor characteristics of participants in Phase 2a

  1. Cohort A: Tumor p53 wild-type with histologically confirmed diagnosis of advanced or metastatic DD LPS (and MDM2 amplification); OR Cohort B: Tumor p53 wild-type in other solid tumor.
  2. Measurable disease by RECIST 1.1.
* 18 years old or older.
* Resolution of clinically relevant toxicity-related to prior anticancer therapies prior to receipt of study treatment to Grade 1 or less.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants of childbearing/reproductive potential must agree to use adequate birth control measures during the course of the trial and for at least 3 months after discontinuing study treatment.

Exclusion Criteria:

* Anticipated need for major surgery and/or localized palliative radiation within the next 6 weeks
* Active, untreated central nervous system metastases. Participants with brain metastases identified at Screening may be rescreened after the lesion(s) have been appropriately treated; participants with treated brain metastases should be neurologically stable for 4 weeks post-treatment and prior to study enrollment, and off corticosteroids for at least 2 weeks before start of study treatment, and treated lesions should demonstrate no new growth on the re-screening scan.
* Known HIV infection or active hepatitis B or C infection.
* Thrombotic event requiring active and ongoing anticoagulation within the last 6 months prior to study treatment.
* Myocardial infarction within the last 6 months prior to study treatment.
* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension or arrhythmia, congestive heart failure New York Heart Association (NYHA) Class III or IV related to primary cardiac disease, uncontrolled ischemic or severe vascular heart disease.
* A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Known bleeding disorder (e.g., hemophilia, von Willebrand disease).
* Conditions that may predispose to major bleeding (e.g., active GI ulcers, upper or lower GI bleedings in the last 6 months, significant hemoptysis in the last 6 months, tumor invasion of major vessels, etc.). Conditions that have been treated may be allowed if resolution of the risk is documented.
* Use or indication for full dose anticoagulation or anti-platelet therapy including low dose aspirin.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of DLT | 21 days
  Incidence of DLT in Cycle 1 (Day 1 to 21)
Phase 1 and 2: Adverse events | Approximately 2 years
  Frequency of adverse events

SECONDARY OUTCOMES:
Phase 1: Peak plasma concentration | Day 4
  Determine the pharmacokinetic profile of SA53-OS (Cmax)
Phase 1: Area under the plasma concentration versus time curve between 0 and 24 hours | Day 4
  Determine the pharmacokinetic profile of SA53-OS (AUC0-24)
Phase 1: Half-life | Day 4
  Determine the pharmacokinetic profile of SA53-OS (T1/2)
Phase 2: Objective response rate (ORR) | Approximately 2 years
  Participants achieving ORR defined as complete response (CR) rate plus partial response (PR) rate.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Phase 2: Progression free survival (PFS) | Approximately 2 years
  Participants not meeting the definition for progressive disease
Phase 2: Overall survival | Approximately 2 years
  To evaluate overall survival
Phase 2: Duration of response | Approximately 2 years
  Duration of response will be evaluated in responders
Phase 2: Complete response rate | Approximately 2 years
  Participants achieving CR defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Phase 2: Stable disease rate | Approximately 2 years
  Participants achieving stable disease defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Phase 2: Disease control rate | Approximately 2 years
  Participants achieving CR + PR + stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Hanna, MD, Study Director — Lamassu Bio
Locations (2):
- United States (2):
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio